CLINICAL TRIAL: NCT03023345
Title: Evaluation of the Feasibility and Tolerance of Trans-rectal Focal Microwave Ablation of the Index Tumor in Patients With Low-risk Prostate Cancer
Brief Title: Trans-rectal Focal Microwave Ablation of the Index Tumor in Patients With Low-risk Prostate Cancer
Acronym: FOSTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Unité de Recherche Clinique Necker Cochin, Fr (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160301
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Low-Risk Prostate Cancer
Keywords: cancer; prostate; PSA; biopsies; microwave trans rectal focal treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microwave (Experimental): Microwave trans rectal focal treatment
  Interventions: Device: Microwave trans rectal focal treatment

INTERVENTIONS:
Device: Microwave trans rectal focal treatment — Microwave trans-rectal ablation of the prostatic index tumor using MRI-transrectal ultrasound image registration
  Other Names: Microwave thermal ablation system called TATO (Biomedical)

SUMMARY:
The purpose of this study is to determine if trans-rectal microwave ablation of the index tumor of patients with low-risk prostate cancer is sufficiently precise and safe, using MRI-transrectal ultrasound image registration.

DETAILED DESCRIPTION:
In men with low-risk prostate cancer, European and American guidelines recommend either active surveillance or whole-gland treatments, with significant induced morbidity and burden on quality of life. Focal treatments of the index tumor are currently under investigation to decrease morbidity while proposing active treatment.

The purpose of this study is to determine the feasibility, precision and safety of a novel ablation treatment using microwaves, delivered transrectally under real-time guidance with MRI-transrectal ultrasound image registration. The index tumor will be detected with prostate MRI and characterized with targeted biopsies using MRI-transrectal ultrasound image registration. It will then be ablated with microwaves using the same transrectal approach and guidance system (KOELIS).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 45 to 76 years old ;
* Life expectancy above 10 years ;
* Diagnosis of prostate cancer confirmed on prostate biopsies ;
* Low risk of progression, defined with D'Amico criteria :

  * T1c or T2a stage
  * Maximum Gleason score of 3+4, including targeted biopsies corresponding to less than 50% grade 4 for the tumor
  * Prostate Specific Antigen <15 ng/mL
* Detection of the index tumor with prostate MRI, characterized with targeted biopsies using MRI-transrectal ultrasound image registration ;
* Patient accepting to be followed after the procedure using active surveillance protocol standards ;
* Patient affiliated to national health care insurance ;
* Free consent, informed and written, dated and signed by the patient and the investigator before enrollment.

Exclusion Criteria:

* Medical past history of prostatic surgery ;
* Medical past history of radiotherapy or pelvic trauma ;
* Medical past history of acute or chronic prostatitis
* severe BPH-related urinary tract symptoms defined as an IPSS >18 ;
* Extra-capsular extension or seminal vesicle invasion on prostate MRI.
* Tumor involvement > 3 mm on systematic biopsies outside the tumor volume detected on MRI.
* Tumor largest axis > 20 mm on prostate MRI ;
* Distance of less than 5 mm between the tumor and the rectum
* Patient unable to understand the course of the study
* History of allergy or non-tolerance to gadolinium salts used in MRI
* Patient with a contraindication to performing an MRI
* Person placed under safeguard of justice

Ages: 45 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Complete necrosis of the index tumor on prostate MRI | 7 days

SECONDARY OUTCOMES:
Margins of necrosis around the index tumor on prostate MRI | 7 days
Erectile and Ejaculatory function using the International Index Erectile Function (IIEF) self questionnaire | 7 days
  to assess sexual tolerance
Erectile and Ejaculatory function using the International Index Erectile Function (IIEF) self questionnaire | 1 month
  to assess sexual tolerance
Erectile and Ejaculatory function using the International Index Erectile Function (IIEF) self questionnaire | 3 months
  to assess sexual tolerance
Erectile and Ejaculatory function using the International Index Erectile Function (IIEF) self questionnaire | 6 months
  to assess sexual tolerance
Urinary symptoms using IPSS | 7 days
  to assess urinary tolerance
Urinary symptoms using IPSS | 1 month
  to assess urinary tolerance
Urinary symptoms using IPSS | 3 months
  to assess urinary tolerance
Urinary symptoms using IPSS | 6 months
  to assess urinary tolerance
Number of cancer on targeted biopsies within the treated volume | 6 months
  to assess oncological efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BARRY DELONGCHAMPS, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry Delongchamps N, Schull A, Anract J, Abecassis JP, Zerbib M, Sibony M, Jilet L, Abdoul H, Goffin V, Peyromaure M. Feasibility and safety of targeted focal microwave ablation of the index tumor in patients with low to intermediate risk prostate cancer: Results of the FOSTINE trial. PLoS One. 2021 Jul 14;16(7):e0252040. doi: 10.1371/journal.pone.0252040. eCollection 2021. PMID 34260598